CLINICAL TRIAL: NCT06331819
Title: Clinical Association Between Obstructive Sleep Apnea (OSA) and Facial Pigmentation, and the Relation Between OSA and Vasovagal Symptoms With Resulting Smoking Tendency and the Effect of Treatment in Patients Referred for Sleep Study.
Brief Title: Clinical Association Between Obstructive Sleep Apnea, Facial Pigmentation, and Vasovagal Symptoms.
Acronym: VasOSA
Status: Recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: 7-3-2024
Record Dates: First submitted 2024-03-07; First posted 2024-03-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea; Vasovagal Syncope; Smoking; Acanthosis Nigricans
Keywords: Obstructive Sleep Apnea; Vasovagal Syncope; Facial Discoloration; Acanthosis Nigricans; Smoking Cessation; Jordan; In-Lab Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Syncope, Vasovagal; Smoking; Acanthosis Nigricans; Smoking Cessation | interventions — Polysomnography; Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients referred for sleep study by in-lab polysomnography to enrolled hospitals and those provided with an at-home sleep study kit.
  Interventions: Diagnostic Test: In-lab polysomnography; Device: Continuous positive airway pressure; Diagnostic Test: Home sleep study device

INTERVENTIONS:
Diagnostic Test: In-lab polysomnography — Patient's brainwaves are recorded overnight to diagnose sleep disorder.
  Other Names: Sleep study
Device: Continuous positive airway pressure — A machine that uses air pressure to keep breathing airways open while patients sleep.
  Other Names: CPAP
Diagnostic Test: Home sleep study device — Patient's brainwaves are recorded overnight to diagnose sleep disorder.

SUMMARY:
The goal of this prospective cohort study is to study patients referred for sleep study by in-lab polysomnography in the Jordan University Hospital and the Jordan Hospital or with an at-home sleep study kit. The main aims are:

* To prospectively obtain demographic and clinical information of patients referred for a sleep study.
* To determine the diagnostic value of facial discoloration as potential marker for obstructive sleep apnea to increase detection rate for the condition.
* To establish a correlation between obstructive sleep apnea and vasovagal symptoms with resulting increased smoking tendency and study the effect of treatment on the disorders.
* To determine the association between timing of appearance of obstructive sleep apnea symptoms and initiation of smoking.

DETAILED DESCRIPTION:
In this prospective cohort study, participants referred for a sleep study by in-lab polysomnography at the Jordan University Hospital and those who preferred their study conducted at a private clinic or with an at-home sleep study kit will be screened and physically examined for any facial discoloration which will be accordingly graded as low, moderate, or high based on severity of difference from normal skin colour and texture and pictured with patients' consent and privacy maintained. In addition to a general history, participants will be asked in detail about their smoking habits, vasovagal symptoms, sleeping habits, and any specific obstructive sleep apnea symptoms. After the sleep study is performed, positive and negative results will be collected and correlated with presence of facial discolouration. Severity of OSA will be graded by apnea-hypopnea index (AHI) and recorded as mild (5 - 15 events/hour), moderate (15 - 30 events/hour), or severe (> 30 events/hour). Participants with positive results will then be followed up with at 3 weeks and 6 months to determine what treatment they were given, assessed for improvement on treatment, and be questioned regarding smoking and vasovagal symptoms again. Improvement is defined as better sleep quality and reduction of initial symptoms. Participants with negative results will also be followed up with and asked about their smoking habits and vasovagal symptoms. Correlation will then be made between the group that improved on treatment and the group that did not (whether due to ineffective treatment or not receiving treatment at all) to see if improvement reduces smoking tendency with alleviated vasovagal symptoms, and compared with participants with negative sleep study results for any change in smoking habits as well.

A purposive sampling technique will be utilized to determine the study population. The target population is patients above the age of 18 referred for sleep study at the Jordan University Hospital and Jordan Hospital. Patients who agree to participate in this study and sign the consent form.

Researchers will interview patients in person at their initial sleep study visit to physically examine and observe participants' faces for discoloration and take pictures for future reference with consent. Follow up at 3 weeks and 6 months will be done either in the clinic or over the phone and Email.

The data will be analysed using frequencies, means, standard deviations, and chi-square tests using SPSS for windows. The chi-square test will be used to assess the significance of the correlation between obstructive sleep apnea and facial discolouration, which will be considered significant at below p<0.05. Prevalence of vasovagal symptoms as well as smoking habits in patients referred for polysomnography will be recorded and evaluated for significance, and then compared with patients' follow up at 3 weeks and 6 months to assess changes on improvement using the chi-square test as well.

Informed consent will be obtained from participants with anonymity confidentiality assured. The study will be explained to patients, after which they must sign a consent form. Each will be assigned a number and the collected data will be used for analysis without reference to patients' identities. Participation does not add risk to the patients since their treatment plan will not be altered, only followed up with.

ELIGIBILITY:
Inclusion Criteria:

* Patients within age limit who agree to participate and sign the consent form.

Exclusion Criteria:

* Patients with prior diagnosis of obstructive sleep apnea by sleep study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is patients above the age of 18 referred for sleep study at referred hospital. Patients who agree to participate in this study must sign the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical association between obstructive sleep apnea and presence of facial pigmentation | Immediate after sleep study result
  Number of patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study and the presence of pigmentation on the face.
Clinical association between obstructive sleep apnea and severity of facial pigmentation | Immediate after sleep study result
  Grade of facial pigmentation in comparison with normal skin tone as low, moderate, or high in patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study.
Relation between obstructive sleep apnea and vasovagal symptoms | 6 months
  Presence of vasovagal symptoms in patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study.
Relation between obstructive sleep apnea and resulting smoking tendency due to vasovagal symptoms | 6 months
  Frequency of smokers in patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study.

SECONDARY OUTCOMES:
Relation between obstructive sleep apnea and the effect of treatment on facial discolouration | 6 months
  Presence or grade of facial discoloration after patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study receive treatment
Relation between obstructive sleep apnea and the effect of treatment on vasovagal symptoms | 6 months
  Presence of vasovagal symptoms after patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study receive treatment
Relation between obstructive sleep apnea and the effect of treatment on smoking habits | 6 months
  Frequency of smokers after patients with a confirmed diagnosis of OSA by in-lab polysomnography or at-home sleep study receive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rand M Zaqqa, Principal Investigator — Jordan University Hospital
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Bonsignore MR, Saaresranta T, Riha RL. Sex differences in obstructive sleep apnoea. Eur Respir Rev. 2019 Nov 6;28(154):190030. doi: 10.1183/16000617.0030-2019. Print 2019 Dec 31. PMID 31694839
- [Background] Eckert DJ, Malhotra A, Jordan AS. Mechanisms of apnea. Prog Cardiovasc Dis. 2009 Jan-Feb;51(4):313-23. doi: 10.1016/j.pcad.2008.02.003. PMID 19110133
- [Background] White DP. Pathogenesis of obstructive and central sleep apnea. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1363-70. doi: 10.1164/rccm.200412-1631SO. Epub 2005 Aug 11. PMID 16100008
- [Background] Green ME, Bernet V, Cheung J. Thyroid Dysfunction and Sleep Disorders. Front Endocrinol (Lausanne). 2021 Aug 24;12:725829. doi: 10.3389/fendo.2021.725829. eCollection 2021. PMID 34504473
- [Background] Ioannidou D, Kalamaras G, Kotoulas SC, Pataka A. Smoking and Obstructive Sleep Apnea: Is There An Association between These Cardiometabolic Risk Factors?-Gender Analysis. Medicina (Kaunas). 2021 Oct 20;57(11):1137. doi: 10.3390/medicina57111137. PMID 34833356
- [Background] Schrand JR. Is sleep apnea a predisposing factor for tobacco use? Med Hypotheses. 1996 Dec;47(6):443-8. doi: 10.1016/s0306-9877(96)90155-3. PMID 8961240
- [Background] Gozal D, Ham SA, Mokhlesi B. Sleep Apnea and Cancer: Analysis of a Nationwide Population Sample. Sleep. 2016 Aug 1;39(8):1493-500. doi: 10.5665/sleep.6004. PMID 27166241
- [Background] Soundararajan V, Lor J, Fishbein AB. Sleep Apnea and Skin. Curr Sleep Med Rep. 2020 Sep;6(3):94-100. doi: 10.1007/s40675-020-00179-7. Epub 2020 Aug 25. PMID 33767945
- [Background] Tien KJ, Chou CW, Lee SY, Yeh NC, Yang CY, Yen FC, Wang JJ, Weng SF. Obstructive sleep apnea and the risk of atopic dermatitis: a population-based case control study. PLoS One. 2014 Feb 25;9(2):e89656. doi: 10.1371/journal.pone.0089656. eCollection 2014. PMID 24586942
- [Background] Jeanmonod R, Sahni D, Silberman M. Vasovagal Episode. 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470277/ PMID 29262088
- [Background] Puel V, Pepin JL, Gosse P. Sleep related breathing disorders and vasovagal syncope, a possible causal link? Int J Cardiol. 2013 Sep 30;168(2):1666-7. doi: 10.1016/j.ijcard.2013.03.061. Epub 2013 Apr 23. No abstract available. PMID 23623670
- [Background] Willis FB, Isley AL, Geda YE, Shaygan A, Quarles L 4th, Fredrickson PA. Resolution of syncope with treatment of sleep apnea. J Am Board Fam Med. 2008 Sep-Oct;21(5):466-8. doi: 10.3122/jabfm.2008.05.070274. PMID 18772302
- [Background] Tayade MC, Kulkarni NB. The effect of smoking on the cardiovascular autonomic functions: a cross sectional study. J Clin Diagn Res. 2013 Jul;7(7):1307-10. doi: 10.7860/JCDR/2013/5526.3133. Epub 2013 Jul 1. PMID 23998052

DOCUMENTS (1):
  • Study Protocol (2024-09-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06331819/Prot_001.pdf